CLINICAL TRIAL: NCT00976040
Title: A Randomized Clinical Trial of Immediate Versus Standard Antiretroviral Therapy for HIV-infected Adults Presenting With Cryptococcal Meningitis
Brief Title: Optimal Time to Start Antiretroviral Therapy in HIV-infected Adults With Cryptococcal Meningitis
Acronym: Crypto
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Botswana-UPenn Partnership (Other)
Collaborators: Doris Duke Charitable Foundation (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Gregory Bisson, Assistant Professor of Medicine, Botswana-UPenn Partnership
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THE BOTSHELO STUDY
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Cryptococcal Meningitis; HIV Infections
Keywords: HIV-1; Africa; Botswana; Highly active antiretroviral therapy; treatment naive
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early antiretroviral therapy (Experimental): Subjects randomized to this arm will initiate antiretroviral therapy within 7 days of enrollment.
  Interventions: Other: Early antiretroviral therapy
- Standard antiretroviral therapy (No Intervention): Subjects randomized to this arm will initiate antiretroviral therapy approximately 4 weeks after enrollment.

INTERVENTIONS:
Other: Early antiretroviral therapy — The intervention is early initiation of antiretroviral therapy after diagnosis of Cryptococcal meningitis.
  In the intervention/experimental arm, triple-drug highly active antiretroviral therapy regimens will be initiated within 7 days of diagnosis of Cryptococcal meningitis.
  Arms: Early antiretroviral therapy

SUMMARY:
The goal of this randomized clinical trial is to compare early versus standard timing of initiation of antiretroviral therapy (ART) with respect to clearance of Cryptococcus neoformans from cerebrospinal fluid (CSF) among HIV-infected adults with Cryptococcal Meningitis.

The investigators hypothesize that early ART mediates more rapid clearance of C. neoformans from CSF, as manifested by a greater rate of decrease in C. neoformans colony forming units (CFUs) during the first 28 days after initiating antifungal treatment.

Secondary hypotheses are that recovery of pathogen specific cellular immunity directed at C. neoformans, as manifested by increases in the number and function of C. neoformans-specific peripheral blood mononuclear cells is associated with 1) ART and 2) pathogen clearance. In addition, patients randomized to the intervention arm will have more rapid clearance of antigen levels in CSF and serum and will have a lower incidence of grade 3 and 4 Adverse events.

ELIGIBILITY:
Inclusion Criteria:

* HIV 1 infection confirmed by licensed ELISA kit and/or detectable Viral load.
* Confirmed Cryptococcal meningitis on the current admission by India ink or CSF cryptococcal antigen
* ART naive at the time of enrollment
* 21 years old and above
* Ability and willingness to give written informed consent to participate in the study
* Able (as assessed by the patient's medical team)to initiate amphotericin B for cryptococcal meningitis
* Initiated amphotericin B 72 hours or less prior to assessment for enrollment or not on amphotericin B at the time of assessment for enrollment
* Agrees to obtain outpatient care after discharge within 50 kilometers from Princess Marina Hospital,Scottish Livingstone Hospital and Bamalete Lutheran Hospital

Exclusion Criteria:

* Recent (within the past 4 weeks) antifungal use
* Pregnant or breastfeeding
* Initiated anti-tubercular therapy 2 weeks or less prior to assessment for enrollment.
* Bacterial meningitis at the time of assessment for enrollment.
* Recent (within the past 1 month) use of the following:systemic cancer chemotherapy,oral or intravenous corticosteroids or other immunomodulators.
* Judged by study coordinator to be likely to initiate chemotherapy or any other immunomodulatory therapy prior to the 4 week LP.
* Imprisoned.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in the CSF CFUs between the immediate and standard ART initiation groups | 4 weeks

SECONDARY OUTCOMES:
Grade 3 or 4 adverse events | 6 months
  each participant is followed up for 6 months after the initiation of HAART
Clearance of C. neoformans antigen from CSF and blood. | 6 months
Change in the number of peripheral blood mononuclear cells responding to C. neoformans | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Bisson, MD,MSCE, Principal Investigator — Botswana-UPenn Partnership, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania; Pablo Tebas, MD, Principal Investigator — Botswana-UPenn Partnership, University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
Locations (1):
- Princess Marina Hospital,Bamalete Lutheran Hospital and Scottish Livingstone Hospital, Gaborone,Ramotswa,Molepolole, Botswana

REFERENCES:
- [Derived] Bisson GP, Molefi M, Bellamy S, Thakur R, Steenhoff A, Tamuhla N, Rantleru T, Tsimako I, Gluckman S, Ravimohan S, Weissman D, Tebas P. Early versus delayed antiretroviral therapy and cerebrospinal fluid fungal clearance in adults with HIV and cryptococcal meningitis. Clin Infect Dis. 2013 Apr;56(8):1165-73. doi: 10.1093/cid/cit019. Epub 2013 Jan 29. PMID 23362285